CLINICAL TRIAL: NCT02006823
Title: Patient Self-management and Gene Guided Therapy for Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00035949
Record Dates: First submitted 2013-11-22; First posted 2013-12-10 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will explore ways to improve the effectiveness of patient Self Management at a time when genetic test results guide new treatments that will dramatically increase the possibility of cure of the hepatitis C virus.The study will also focus on the interactions between provider and patients and the ways that technical work, adaptive work and adaptive leadership foster patient self-management.This proposed 2 year exploratory mixed-methods 12 longitudinal case study will explore patients' and providers' explanations for how and why they engage in technical work, adaptive work, and adaptive leadership and the ways in which these strategies promote or pose barriers to patients' self-management of Chronic Hepatitis C in the context of the new genetic test results and treatments. Specific aims are to:

1: Examine how technical work, adaptive work and adaptive leadership influence patients' perceptions of their likelihood of cure and how this work relates to self-management during 12 to 24 weeks of treatment for Chronic Hepatitis C. Research questions are: 1.1) How do patients describe their interactions with the providers? 1.2) How do these interactions shape patients' perceptions of the likelihood of cure? 1.3) How do patients' understanding of their interactions with the provider promote the use of or pose barriers to self-management during treatment?

AIM 2: Describe providers' use of technical work, and adaptive leadership approaches during clinical encounters,to include nurse education visits. Research questions are:

2.1) What technical work, and adaptive leadership approaches do providers use when sharing treatment information with patients during the clinical encounters. 2.2) What explanations do providers give for how and why they use technical work and adaptive leadership approaches? AIM 3: Describe the trajectories of illness perceptions(Control/Cure sub-scale - Illness Perception Scale), symptoms (M.D. Anderson Symptom Inventory) , viral load, and self-management (Patient Activation Measure) in relation to patient and provider reports of technical work, adaptive work, and adaptive leadership from the index clinical encounter to the follow-up treatment response encounter (ranging from 12 to 24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* African American or Caucasian
* Genotype 1
* Planning to, but have not yet, began treatment for Hepatitis C at Duke University Medical Center or Boice-Willis Clinic in Rocky Mount, NC

Exclusion Criteria:

* Diagnosed with Bipolar Disorder or Schizophrenia
* Not genotype 1
* Any race other than African American or Caucasian.
* Hispanic or Latino

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African-American or Caucasian patients with Type 1 Chronic Hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in Self Management | baseline, 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks, 18 weeks, 24 weeks
  Self Management as measured by the Patient Activation Measure which is an measure of their responses. The study team will plot a trajectory line using the Patient Activation Measure across all time points. The team is interested in knowing if this measure changes based on the patients self-management and his/her interaction with the health care provider.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Bailey, PhD, Principal Investigator — Duke University School of Nursing
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Boice Willis Clinic, Rocky Mount, North Carolina

REFERENCES:
- [Derived] Bailey DE Jr, Hendrix CC, Steinhauser KE, Stechuchak KM, Porter LS, Hudson J, Olsen MK, Muir A, Lowman S, DiMartini A, Salonen LW, Tulsky JA. Randomized trial of an uncertainty self-management telephone intervention for patients awaiting liver transplant. Patient Educ Couns. 2017 Mar;100(3):509-517. doi: 10.1016/j.pec.2016.10.017. Epub 2016 Oct 18. PMID 28277289